CLINICAL TRIAL: NCT02914405
Title: A Phase I Study of 131-1 mIBG Followed by Nivolumab and Dinutuximab Beta in Children With Relapsed/Refractory Neuroblastoma
Brief Title: Phase I Study of 131-I mIBG Followed by Nivolumab & Dinutuximab Beta Antibodies in Children With Relapsed/Refractory Neuroblastoma
Acronym: MiniVan
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: University College London Hospitals (Other); University of Wisconsin, Madison (Other); University Hospital Greifswald (Other); Solving Kids' Cancer US/EU (Unknown); Joining Against Cancer in Kids (Unknown); The Band of Parents (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RHM CHI0811; 2016-002221-11 (EudraCT Number)
Record Dates: First submitted 2016-08-25; First posted 2016-09-26 (Estimated); Last update posted 2025-10-22 (Actual); Status verified 2024-12

CONDITIONS: Neuroblastoma
Keywords: 131-I-mIBG therapy; ch14.18/CHO; Nivolumab; MiniVan
MeSH Terms: conditions — Neuroblastoma | interventions — Nivolumab; Immunoglobulin G; Antibodies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Experimental): The dose and schedule of 131-I mIBG will be constant, and the doses of ch14.18/ CHO and Nivolumab determined by cohort:
  * Cohort I: 3 mg/kg Nivolumab (100% adult dose). No ch14.18/CHO. (3-6 patients)
  * Cohort II: 50mg/m2/cycle ch14.18/CHO (50% established Long Term Intervention (LTI) dose) and 3 mg/kg Nivolumab (100% adult dose) (3-6 patients)
  * Cohort III: 100mg/m2/cycle ch14.18/CHO (100% established LTI dose) and 3 mg/kg Nivolumab (100% adult dose) (initial 3-6 patients, expanded to 15 patient cohort if tolerated)
  Interventions: Drug: Nivolumab; Drug: Ch14.18/CHO

INTERVENTIONS:
Drug: Nivolumab — Nivolumab is a soluble protein consisting of 4 polypeptide chains, which include 2 identical heavy chains consisting of 440 amino acids and 2 identical light chains. Molecular weight is 146,221 daltons.
  Other Names: BMS-936558; MDX1106; ONO-4538; anti-PD-1) NSC#748726; IND #124729
Drug: Ch14.18/CHO — APN311 (ch14.18/CHO) is manufactured in a Good Manufacturing Practice (GMP) compliant facility of Polymun Scientific, Austria according to a state of the art aseptic manufacturing process based on a characterized and stable Chinese Hamster Ovary (CHO) cell line. After propagation of the working cell bank (WCB) in small volume vessels/bioreactors, manufacture is carried out in a 2500 L stirred tank reactor utilizing components which are free of material of animal or human origin.
  Other Names: Mouse-human chimeric monoclonal anti-GD2 Immunoglobulin G1 (IgG1) antibody

SUMMARY:
Neuroblastoma, the most common extra-cranial solid tumour in children, remains one of the major challenges in paediatric oncology. A promising way to further improve outcome in this disease appears to be the development of adjuvant therapeutic strategies. In this research the anti-GD2 antibody, which is a standard treatment, is to be combined with 131-l Metaiodobenzylguanidine (mlBG) and anti-Programmed Cell Death Protein 1 (anti-PD1) antibody Nivolumab - the investigated drugs - with the aim of generating sustained anti-neuroblastoma immunity. In particular it will be determined the safety and tolerability of the novel combination as well as documented any evidence of efficacy in paediatric patients with relapsed and refractory high risk neuroblastoma.

This study is sponsored by the University Hospital Southampton and will take place in 4 hospitals in the United Kingdom, Germany and USA. The estimated duration of the study is 2 years, starting in December 2016.

This is an "adaptive study". Such design uses accumulating of data from the ongoing trial to modify aspects of the study (e.g. duration, number of treatments) without undermining its validity or integrity. There will be 3 cohorts of patients. As safety of Nivolumab is well established, Cohort 1 will assess its safety and tolerability in combination with 131-l mlBG. Cohort 2 will then add anti-GD2 to the drug combination, assessing safety and tolerability. Cohort 3 will escalate all 3 agents to the full 100% dose level to assure safety for expanded analyses of clinical and laboratory data at that dose level.

Patients will initially be recruited into Cohort 1. Patients must have completed at least 12 weeks of trial treatment without reaching a Dose Limiting Toxicity before a patient can be recruited to the next cohort.

A minimum of 3 evaluable patients will be treated in cohorts 1-3. Assuming the full dose combination therapy (cohort) is tolerable, 15 evaluable patients will be treated.

ELIGIBILITY:
Inclusion Criteria:

* At study entry patients must be > 1 year
* Relapsed or refractory high risk neuroblastoma (as defined by International Neuroblastoma Risk Group (INRG) criteria)
* MIBG avid disease on imaging within 4 weeks to study entry.
* ≥ 3 months since any myeloablative chemotherapy / stem cell rescue
* ≥ 42 days since any other immunotherapy e.g. tumour vaccines. At least 3 half lives since last dose of any monoclonal antibody therapy.
* Patients must have a performance status greater or equal 60% (Lansky Score or Karnofsky)
* Estimated life expectancy ≥ 12 weeks
* Adequate bone marrow function: Absolute Neutrophil Count (ANC) >1.0 x 10/L, platelets, 20 x 10/L and haemoglobin > 8.0 g/dL.
* Adequate renal function: serum creatinine <1.5 mg/dL or a estimated creatinine clearance or radioisotope Glomerular Filtration Rate Study (GFR) of > 60 mL/minute/1.73m2.
* Adequate cardiac function: shortening fraction of 28 % by echocardiogram.
* Adequate hepatic function: Alanine transaminase (ALT) or Aspartate transaminase (AST) < 5 x ULN and a total bilirubin < 1.5 x Upper Limit of Normal (ULN)
* Adequate lung function: Forced Expiratory Volume in 1 Second (FEV1) and Forced Vital Capacity (FVC) >60% of the predicted by pulmonary function tests. Children unable to do Pulmonary Function Tests (PFTs) should have no dyspnea at rest and a pulse oximetry >94% on room air.
* Adequate pancreatic function: serum lipase < 1.5 x upper limit normal
* Patients may have had prior Central Nervous System (CNS) metastasis at point of entry to study, but patients with mIBG avid parenchymal brain lesions will be excluded. All CNS disease must be treated and stable prior for at least 4 weeks prior to starting trial 131-I mIBG therapy (see section 4). Patients with extra-axial disease (e.g. skull (bone) metastasis that do not invade the dura) may be enrolled providing there is no evidence of brain oedema.
* Patients must consent to the placement of a central venous line, if one has not already been placed.
* Patients must have no immediate requirements for palliative chemotherapy, radiotherapy or surgery.
* Females of childbearing potential must have a negative pregnancy test. Patients of childbearing potential must agree to use an effective birth control method. Female patients who are lactating must agree to stop breast-feeding.
* Patients with seizure disorders may be enrolled if seizures are well controlled.
* All patients and/or their parents or legal guardians must sign a written informed consent
* All institutional and national requirements for clinical trials must be met.
* Expression of PD-L1 by tumour is not a pre-requisite
* Parents or carers willing and able to comply with radiation safety measures needed for 131-I mIBG administration.
* Patient must be judged capable of tolerating isolation procedures associated with 131-I-mIBG therapy

Exclusion Criteria

* Patients who have previously received ch14.18 (CHO or SP2/0) will not be excluded unless they have had severe or life threatening toxicity necessitating withdrawal of treatment previously or if they have a strong/neutralizing Human Antichimeric Antibody (HACA) (≥ 10 μg/ml)
* Patients who have had previous 131-I mIBG therapy will not be excluded
* Patients previously treated with Nivolumab or any other PD-1 or PD-L1 targeting antibodies will be excluded from the study
* Previous allogeneic stem cell transplant or solid organ transplant
* Patients should be excluded if they have an active, known or suspected autoimmune disease. Subjects are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger
* Patients receiving systemic corticosteroids (other than physiological replacement) or other immunosuppressive agents within 14 days prior to study entry
* Unable to maintain platelets ≥ 50 x 109/l without transfusion
* HIV or Hepatitis B or C infection
* Patients with significant intercurrent illnesses and/or any of the following:

  * Patients with symptoms of congestive heart failure or uncontrolled cardiac rhythm disturbance.
  * Patients with significant psychiatric disabilities or uncontrolled seizure disorders.
  * Patients with active infections.
  * Patients with a clinically significant neurologic deficit or objective peripheral neuropathy (Grade >2) are ineligible.
  * Patients with clinically significant, symptomatic, pleural effusions.
  * Patients who require, or are likely to require, corticosteroid or other immunosuppressive drugs.

Ages: 1 Year to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2018-05-24 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and tolerability] of 131-I-MIBG, ch14.18/CHO and Nivolumab in paediatric patients | 2 Years
  • To determine the safety and tolerability of the novel combination of 131-I-MIBG, ch14.18/CHO and Nivolumab in paediatric patients, assessed by nature, frequency, severity and timing of adverse events, including serious adverse events and immune related adverse events during administration of ch14.18/CHO

SECONDARY OUTCOMES:
Anti-tumour response in patients with measureable disease as measured by immunocytology, MIBG, CT and/or MRI in patients receiving 131-I-MIBG, ch14.18/CHO and Nivolumab in patients with relapsed and refractory high risk neuroblastoma | 2 Years
  To document any evidence of efficacy of 131-I-MIBG, ch14.18/CHO and Nivolumab in patients with relapsed and refractory high risk neuroblastoma (time to progression)
Anti-tumour response in patients with measureable disease as measured by immunocytology, MIBG, CT and/or MRI in patients receiving 131-I-MIBG, ch14.18/CHO and Nivolumab in patients with relapsed and refractory high risk neuroblastoma | 2 Years
  To document any evidence of efficacy of 131-I-MIBG, ch14.18/CHO and Nivolumab in patients with relapsed and refractory high risk neuroblastoma (objective response rate)
KIR/KIR-Ligand genotype, FcγR genotype | 2 Years
  To provide descriptive analysis of any associations between KIR/KIR-Ligand genotype, FcγR genotype and response

CONTACTS AND LOCATIONS:
Overall Officials: Juliet Gray, Principal Investigator — Consultant Paediatric Oncologist
Locations (3):
- University of Wisconsin Carbone Cancer Center; UW Hospital and Clinics; American Family Children's Hospital, Madison, Wisconsin, United States
- United Kingdom (2):
  - University Hospital Southampton NHS Foundation Trust, Southampton, Hampshire
  - University College London Hospital, London, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garra G, Singer AJ, Taira BR, Chohan J, Cardoz H, Chisena E, Thode HC Jr. Validation of the Wong-Baker FACES Pain Rating Scale in pediatric emergency department patients. Acad Emerg Med. 2010 Jan;17(1):50-4. doi: 10.1111/j.1553-2712.2009.00620.x. Epub 2009 Dec 9. PMID 20003121
- [Background] Hicks CL, von Baeyer CL, Spafford PA, van Korlaar I, Goodenough B. The Faces Pain Scale-Revised: toward a common metric in pediatric pain measurement. Pain. 2001 Aug;93(2):173-183. doi: 10.1016/S0304-3959(01)00314-1. PMID 11427329
- [Background] Bulloch B, Tenenbein M. Validation of 2 pain scales for use in the pediatric emergency department. Pediatrics. 2002 Sep;110(3):e33. doi: 10.1542/peds.110.3.e33. PMID 12205283
- [Background] Wilson GA, Doyle E. Validation of three paediatric pain scores for use by parents. Anaesthesia. 1996 Nov;51(11):1005-7. doi: 10.1111/j.1365-2044.1996.tb14991.x. PMID 8943588
- [Background] Buttner W, Breitkopf L, Miele B, Finke W. [Initial results of the reliability and validity of a German-language scale for the quantitative measurement of postoperative pain in young children]. Anaesthesist. 1990 Nov;39(11):593-602. German. PMID 2288408
- [Background] Ramsay MA, Savege TM, Simpson BR, Goodwin R. Controlled sedation with alphaxalone-alphadolone. Br Med J. 1974 Jun 22;2(5920):656-9. doi: 10.1136/bmj.2.5920.656. PMID 4835444
- [Result] Matthay KK, Yanik G, Messina J, Quach A, Huberty J, Cheng SC, Veatch J, Goldsby R, Brophy P, Kersun LS, Hawkins RA, Maris JM. Phase II study on the effect of disease sites, age, and prior therapy on response to iodine-131-metaiodobenzylguanidine therapy in refractory neuroblastoma. J Clin Oncol. 2007 Mar 20;25(9):1054-60. doi: 10.1200/JCO.2006.09.3484. PMID 17369569
- [Result] Matthay KK, Quach A, Huberty J, Franc BL, Hawkins RA, Jackson H, Groshen S, Shusterman S, Yanik G, Veatch J, Brophy P, Villablanca JG, Maris JM. Iodine-131--metaiodobenzylguanidine double infusion with autologous stem-cell rescue for neuroblastoma: a new approaches to neuroblastoma therapy phase I study. J Clin Oncol. 2009 Mar 1;27(7):1020-5. doi: 10.1200/JCO.2007.15.7628. Epub 2009 Jan 26. PMID 19171714
- [Result] Matthay KK, Weiss B, Villablanca JG, Maris JM, Yanik GA, Dubois SG, Stubbs J, Groshen S, Tsao-Wei D, Hawkins R, Jackson H, Goodarzian F, Daldrup-Link H, Panigrahy A, Towbin A, Shimada H, Barrett J, Lafrance N, Babich J. Dose escalation study of no-carrier-added 131I-metaiodobenzylguanidine for relapsed or refractory neuroblastoma: new approaches to neuroblastoma therapy consortium trial. J Nucl Med. 2012 Jul;53(7):1155-63. doi: 10.2967/jnumed.111.098624. Epub 2012 Jun 14. PMID 22700000
- [Result] Wilson JS, Gains JE, Moroz V, Wheatley K, Gaze MN. A systematic review of 131I-meta iodobenzylguanidine molecular radiotherapy for neuroblastoma. Eur J Cancer. 2014 Mar;50(4):801-15. doi: 10.1016/j.ejca.2013.11.016. Epub 2013 Dec 12. PMID 24333097
- [Result] Gaze MN, Chang YC, Flux GD, Mairs RJ, Saran FH, Meller ST. Feasibility of dosimetry-based high-dose 131I-meta-iodobenzylguanidine with topotecan as a radiosensitizer in children with metastatic neuroblastoma. Cancer Biother Radiopharm. 2005 Apr;20(2):195-9. doi: 10.1089/cbr.2005.20.195. PMID 15869455
- [Result] Suzuki M, Cheung NK. Disialoganglioside GD2 as a therapeutic target for human diseases. Expert Opin Ther Targets. 2015 Mar;19(3):349-62. doi: 10.1517/14728222.2014.986459. Epub 2015 Jan 20. PMID 25604432
- [Result] Honsik CJ, Jung G, Reisfeld RA. Lymphokine-activated killer cells targeted by monoclonal antibodies to the disialogangliosides GD2 and GD3 specifically lyse human tumor cells of neuroectodermal origin. Proc Natl Acad Sci U S A. 1986 Oct;83(20):7893-7. doi: 10.1073/pnas.83.20.7893. PMID 3094017
- [Result] Gillies SD, Lo KM, Wesolowski J. High-level expression of chimeric antibodies using adapted cDNA variable region cassettes. J Immunol Methods. 1989 Dec 20;125(1-2):191-202. doi: 10.1016/0022-1759(89)90093-8. PMID 2514231
- [Result] Zeng Y, Fest S, Kunert R, Katinger H, Pistoia V, Michon J, Lewis G, Ladenstein R, Lode HN. Anti-neuroblastoma effect of ch14.18 antibody produced in CHO cells is mediated by NK-cells in mice. Mol Immunol. 2005 Jul;42(11):1311-9. doi: 10.1016/j.molimm.2004.12.018. Epub 2005 Apr 7. PMID 15950727
- [Result] Yu AL, Gilman AL, Ozkaynak MF, London WB, Kreissman SG, Chen HX, Smith M, Anderson B, Villablanca JG, Matthay KK, Shimada H, Grupp SA, Seeger R, Reynolds CP, Buxton A, Reisfeld RA, Gillies SD, Cohn SL, Maris JM, Sondel PM; Children's Oncology Group. Anti-GD2 antibody with GM-CSF, interleukin-2, and isotretinoin for neuroblastoma. N Engl J Med. 2010 Sep 30;363(14):1324-34. doi: 10.1056/NEJMoa0911123. PMID 20879881
- [Result] Ora I, Eggert A. Progress in treatment and risk stratification of neuroblastoma: impact on future clinical and basic research. Semin Cancer Biol. 2011 Oct;21(4):217-28. doi: 10.1016/j.semcancer.2011.07.002. Epub 2011 Jul 20. PMID 21798350
- [Result] Handgretinger R, Baader P, Dopfer R, Klingebiel T, Reuland P, Treuner J, Reisfeld RA, Niethammer D. A phase I study of neuroblastoma with the anti-ganglioside GD2 antibody 14.G2a. Cancer Immunol Immunother. 1992;35(3):199-204. doi: 10.1007/BF01756188. PMID 1638557
- [Result] Weiner LM, Dhodapkar MV, Ferrone S. Monoclonal antibodies for cancer immunotherapy. Lancet. 2009 Mar 21;373(9668):1033-40. doi: 10.1016/S0140-6736(09)60251-8. PMID 19304016
- [Result] Saleh MN, Khazaeli MB, Wheeler RH, Dropcho E, Liu T, Urist M, Miller DM, Lawson S, Dixon P, Russell CH, et al. Phase I trial of the murine monoclonal anti-GD2 antibody 14G2a in metastatic melanoma. Cancer Res. 1992 Aug 15;52(16):4342-7. PMID 1643631
- [Result] Murray JL, Cunningham JE, Brewer H, Mujoo K, Zukiwski AA, Podoloff DA, Kasi LP, Bhadkamkar V, Fritsche HA, Benjamin RS, et al. Phase I trial of murine monoclonal antibody 14G2a administered by prolonged intravenous infusion in patients with neuroectodermal tumors. J Clin Oncol. 1994 Jan;12(1):184-93. doi: 10.1200/JCO.1994.12.1.184. PMID 8270976
- [Result] Uttenreuther-Fischer MM, Huang CS, Yu AL. Pharmacokinetics of human-mouse chimeric anti-GD2 mAb ch14.18 in a phase I trial in neuroblastoma patients. Cancer Immunol Immunother. 1995 Dec;41(6):331-8. doi: 10.1007/BF01526552. PMID 8635190
- [Result] Frost JD, Hank JA, Reaman GH, Frierdich S, Seeger RC, Gan J, Anderson PM, Ettinger LJ, Cairo MS, Blazar BR, Krailo MD, Matthay KK, Reisfeld RA, Sondel PM. A phase I/IB trial of murine monoclonal anti-GD2 antibody 14.G2a plus interleukin-2 in children with refractory neuroblastoma: a report of the Children's Cancer Group. Cancer. 1997 Jul 15;80(2):317-33. doi: 10.1002/(sici)1097-0142(19970715)80:23.0.co;2-w. PMID 9217046
- [Result] Saleh MN, Khazaeli MB, Wheeler RH, Allen L, Tilden AB, Grizzle W, Reisfeld RA, Yu AL, Gillies SD, LoBuglio AF. Phase I trial of the chimeric anti-GD2 monoclonal antibody ch14.18 in patients with malignant melanoma. Hum Antibodies Hybridomas. 1992 Jan;3(1):19-24. PMID 1576319
- [Result] Handgretinger R, Anderson K, Lang P, Dopfer R, Klingebiel T, Schrappe M, Reuland P, Gillies SD, Reisfeld RA, Neithammer D. A phase I study of human/mouse chimeric antiganglioside GD2 antibody ch14.18 in patients with neuroblastoma. Eur J Cancer. 1995;31A(2):261-7. doi: 10.1016/0959-8049(94)00413-y. PMID 7718335
- [Result] Yu AL, Uttenreuther-Fischer MM, Huang CS, Tsui CC, Gillies SD, Reisfeld RA, Kung FH. Phase I trial of a human-mouse chimeric anti-disialoganglioside monoclonal antibody ch14.18 in patients with refractory neuroblastoma and osteosarcoma. J Clin Oncol. 1998 Jun;16(6):2169-80. doi: 10.1200/JCO.1998.16.6.2169. PMID 9626218
- [Result] Simon T, Berthold F, Borkhardt A, Kremens B, De Carolis B, Hero B. Treatment and outcomes of patients with relapsed, high-risk neuroblastoma: results of German trials. Pediatr Blood Cancer. 2011 Apr;56(4):578-83. doi: 10.1002/pbc.22693. Epub 2010 Dec 9. PMID 21298742
- [Result] Murray JL, Kleinerman ES, Jia SF, Rosenblum MG, Eton O, Buzaid A, Legha S, Ross MI, Thompson L, Mujoo K, Rieger PT, Saleh M, Khazaeli MB, Vadhan-Raj S. Phase Ia/Ib trial of anti-GD2 chimeric monoclonal antibody 14.18 (ch14.18) and recombinant human granulocyte-macrophage colony-stimulating factor (rhGM-CSF) in metastatic melanoma. J Immunother Emphasis Tumor Immunol. 1996 May;19(3):206-17. doi: 10.1097/00002371-199605000-00005. PMID 8811495
- [Result] Albertini MR, Hank JA, Schiller JH, Khorsand M, Borchert AA, Gan J, Bechhofer R, Storer B, Reisfeld RA, Sondel PM. Phase IB trial of chimeric antidisialoganglioside antibody plus interleukin 2 for melanoma patients. Clin Cancer Res. 1997 Aug;3(8):1277-88. PMID 9815810
- [Result] Ozkaynak MF, Sondel PM, Krailo MD, Gan J, Javorsky B, Reisfeld RA, Matthay KK, Reaman GH, Seeger RC. Phase I study of chimeric human/murine anti-ganglioside G(D2) monoclonal antibody (ch14.18) with granulocyte-macrophage colony-stimulating factor in children with neuroblastoma immediately after hematopoietic stem-cell transplantation: a Children's Cancer Group Study. J Clin Oncol. 2000 Dec 15;18(24):4077-85. doi: 10.1200/JCO.2000.18.24.4077. PMID 11118469
- [Result] Gilman AL, Ozkaynak MF, Matthay KK, Krailo M, Yu AL, Gan J, Sternberg A, Hank JA, Seeger R, Reaman GH, Sondel PM. Phase I study of ch14.18 with granulocyte-macrophage colony-stimulating factor and interleukin-2 in children with neuroblastoma after autologous bone marrow transplantation or stem-cell rescue: a report from the Children's Oncology Group. J Clin Oncol. 2009 Jan 1;27(1):85-91. doi: 10.1200/JCO.2006.10.3564. Epub 2008 Dec 1. PMID 19047298
- [Result] Ladenstein R, Potschger U, Siabalis D, Garaventa A, Bergeron C, Lewis IJ, Stein J, Kohler J, Shaw PJ, Holter W, Pistoia V, Michon J. Dose finding study for the use of subcutaneous recombinant interleukin-2 to augment natural killer cell numbers in an outpatient setting for stage 4 neuroblastoma after megatherapy and autologous stem-cell reinfusion. J Clin Oncol. 2011 Feb 1;29(4):441-8. doi: 10.1200/JCO.2009.23.5465. Epub 2010 Dec 13. PMID 21149662
- [Result] Siebert N, Eger C, Seidel D, Juttner M, Zumpe M, Wegner D, Kietz S, Ehlert K, Veal GJ, Siegmund W, Weiss M, Loibner H, Ladenstein R, Lode HN. Pharmacokinetics and pharmacodynamics of ch14.18/CHO in relapsed/refractory high-risk neuroblastoma patients treated by long-term infusion in combination with IL-2. MAbs. 2016;8(3):604-16. doi: 10.1080/19420862.2015.1130196. Epub 2016 Jan 19. PMID 26785755
- [Result] Weber J. Immune checkpoint proteins: a new therapeutic paradigm for cancer--preclinical background: CTLA-4 and PD-1 blockade. Semin Oncol. 2010 Oct;37(5):430-9. doi: 10.1053/j.seminoncol.2010.09.005. PMID 21074057
- [Result] Callahan MK, Wolchok JD. Clinical Activity, Toxicity, Biomarkers, and Future Development of CTLA-4 Checkpoint Antagonists. Semin Oncol. 2015 Aug;42(4):573-86. doi: 10.1053/j.seminoncol.2015.05.008. Epub 2015 Jun 3. PMID 26320062
- [Result] Barber DL, Wherry EJ, Masopust D, Zhu B, Allison JP, Sharpe AH, Freeman GJ, Ahmed R. Restoring function in exhausted CD8 T cells during chronic viral infection. Nature. 2006 Feb 9;439(7077):682-7. doi: 10.1038/nature04444. Epub 2005 Dec 28. PMID 16382236
- [Result] Dong H, Strome SE, Salomao DR, Tamura H, Hirano F, Flies DB, Roche PC, Lu J, Zhu G, Tamada K, Lennon VA, Celis E, Chen L. Tumor-associated B7-H1 promotes T-cell apoptosis: a potential mechanism of immune evasion. Nat Med. 2002 Aug;8(8):793-800. doi: 10.1038/nm730. Epub 2002 Jun 24. PMID 12091876
- [Result] Iwai Y, Ishida M, Tanaka Y, Okazaki T, Honjo T, Minato N. Involvement of PD-L1 on tumor cells in the escape from host immune system and tumor immunotherapy by PD-L1 blockade. Proc Natl Acad Sci U S A. 2002 Sep 17;99(19):12293-7. doi: 10.1073/pnas.192461099. Epub 2002 Sep 6. PMID 12218188
- [Result] Woo SR, Turnis ME, Goldberg MV, Bankoti J, Selby M, Nirschl CJ, Bettini ML, Gravano DM, Vogel P, Liu CL, Tangsombatvisit S, Grosso JF, Netto G, Smeltzer MP, Chaux A, Utz PJ, Workman CJ, Pardoll DM, Korman AJ, Drake CG, Vignali DA. Immune inhibitory molecules LAG-3 and PD-1 synergistically regulate T-cell function to promote tumoral immune escape. Cancer Res. 2012 Feb 15;72(4):917-27. doi: 10.1158/0008-5472.CAN-11-1620. Epub 2011 Dec 20. PMID 22186141
- [Result] Highfill SL, Cui Y, Giles AJ, Smith JP, Zhang H, Morse E, Kaplan RN, Mackall CL. Disruption of CXCR2-mediated MDSC tumor trafficking enhances anti-PD1 efficacy. Sci Transl Med. 2014 May 21;6(237):237ra67. doi: 10.1126/scitranslmed.3007974. PMID 24848257
- [Result] Zhou Q, Munger ME, Highfill SL, Tolar J, Weigel BJ, Riddle M, Sharpe AH, Vallera DA, Azuma M, Levine BL, June CH, Murphy WJ, Munn DH, Blazar BR. Program death-1 signaling and regulatory T cells collaborate to resist the function of adoptively transferred cytotoxic T lymphocytes in advanced acute myeloid leukemia. Blood. 2010 Oct 7;116(14):2484-93. doi: 10.1182/blood-2010-03-275446. Epub 2010 Jun 22. PMID 20570856
- [Result] Brahmer JR, Tykodi SS, Chow LQ, Hwu WJ, Topalian SL, Hwu P, Drake CG, Camacho LH, Kauh J, Odunsi K, Pitot HC, Hamid O, Bhatia S, Martins R, Eaton K, Chen S, Salay TM, Alaparthy S, Grosso JF, Korman AJ, Parker SM, Agrawal S, Goldberg SM, Pardoll DM, Gupta A, Wigginton JM. Safety and activity of anti-PD-L1 antibody in patients with advanced cancer. N Engl J Med. 2012 Jun 28;366(26):2455-65. doi: 10.1056/NEJMoa1200694. Epub 2012 Jun 2. PMID 22658128
- [Result] Topalian SL, Hodi FS, Brahmer JR, Gettinger SN, Smith DC, McDermott DF, Powderly JD, Carvajal RD, Sosman JA, Atkins MB, Leming PD, Spigel DR, Antonia SJ, Horn L, Drake CG, Pardoll DM, Chen L, Sharfman WH, Anders RA, Taube JM, McMiller TL, Xu H, Korman AJ, Jure-Kunkel M, Agrawal S, McDonald D, Kollia GD, Gupta A, Wigginton JM, Sznol M. Safety, activity, and immune correlates of anti-PD-1 antibody in cancer. N Engl J Med. 2012 Jun 28;366(26):2443-54. doi: 10.1056/NEJMoa1200690. Epub 2012 Jun 2. PMID 22658127
- [Result] Wolchok JD, Kluger H, Callahan MK, Postow MA, Rizvi NA, Lesokhin AM, Segal NH, Ariyan CE, Gordon RA, Reed K, Burke MM, Caldwell A, Kronenberg SA, Agunwamba BU, Zhang X, Lowy I, Inzunza HD, Feely W, Horak CE, Hong Q, Korman AJ, Wigginton JM, Gupta A, Sznol M. Nivolumab plus ipilimumab in advanced melanoma. N Engl J Med. 2013 Jul 11;369(2):122-33. doi: 10.1056/NEJMoa1302369. Epub 2013 Jun 2. PMID 23724867
- [Result] Neal ZC, Yang JC, Rakhmilevich AL, Buhtoiarov IN, Lum HE, Imboden M, Hank JA, Lode HN, Reisfeld RA, Gillies SD, Sondel PM. Enhanced activity of hu14.18-IL2 immunocytokine against murine NXS2 neuroblastoma when combined with interleukin 2 therapy. Clin Cancer Res. 2004 Jul 15;10(14):4839-47. doi: 10.1158/1078-0432.CCR-03-0799. PMID 15269160
- [Result] Lode HN, Xiang R, Varki NM, Dolman CS, Gillies SD, Reisfeld RA. Targeted interleukin-2 therapy for spontaneous neuroblastoma metastases to bone marrow. J Natl Cancer Inst. 1997 Nov 5;89(21):1586-94. doi: 10.1093/jnci/89.21.1586. PMID 9362156
- [Result] Johnson EE, Yamane BH, Buhtoiarov IN, Lum HD, Rakhmilevich AL, Mahvi DM, Gillies SD, Sondel PM. Radiofrequency ablation combined with KS-IL2 immunocytokine (EMD 273066) results in an enhanced antitumor effect against murine colon adenocarcinoma. Clin Cancer Res. 2009 Aug 1;15(15):4875-84. doi: 10.1158/1078-0432.CCR-09-0110. Epub 2009 Jul 28. PMID 19638464
- [Result] Yang RK, Kalogriopoulos NA, Rakhmilevich AL, Ranheim EA, Seo S, Kim K, Alderson KL, Gan J, Reisfeld RA, Gillies SD, Hank JA, Sondel PM. Intratumoral hu14.18-IL-2 (IC) induces local and systemic antitumor effects that involve both activated T and NK cells as well as enhanced IC retention. J Immunol. 2012 Sep 1;189(5):2656-64. doi: 10.4049/jimmunol.1200934. Epub 2012 Jul 27. PMID 22844125
- [Result] Yang RK, Kalogriopoulos NA, Rakhmilevich AL, Ranheim EA, Seo S, Kim K, Alderson KL, Gan J, Reisfeld RA, Gillies SD, Hank JA, Sondel PM. Intratumoral treatment of smaller mouse neuroblastoma tumors with a recombinant protein consisting of IL-2 linked to the hu14.18 antibody increases intratumoral CD8+ T and NK cells and improves survival. Cancer Immunol Immunother. 2013 Aug;62(8):1303-13. doi: 10.1007/s00262-013-1430-x. Epub 2013 May 10. PMID 23661160
- [Result] Williams EL, Dunn SN, James S, Johnson PW, Cragg MS, Glennie MJ, Gray JC. Immunomodulatory monoclonal antibodies combined with peptide vaccination provide potent immunotherapy in an aggressive murine neuroblastoma model. Clin Cancer Res. 2013 Jul 1;19(13):3545-55. doi: 10.1158/1078-0432.CCR-12-3226. Epub 2013 May 6. PMID 23649004
- [Result] Zernikow B, Hechler T. Pain therapy in children and adolescents. Dtsch Arztebl Int. 2008 Jul;105(28-29):511-21; quiz 521-2. doi: 10.3238/arztebl.2008.0511. Epub 2008 Jul 14. PMID 19626208